CLINICAL TRIAL: NCT04118764
Title: Neuronavigation-guided Focused Ultrasound-induced Blood-brain Barrier Opening in Alzheimer's Disease Patients
Brief Title: Non-invasive Blood-brain Barrier Opening in Alzheimer's Disease Patients Using Focused Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAAS5163; R01AG038961 (NIH)
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: focused ultrasound; blood-brain barrier opening; non-invasive therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — perflutren; Magnetic Resonance Spectroscopy; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Focused ultrasound treatment (Experimental): Neuronavigation-guided focused ultrasound treatment in Alzheimer's disease patients using a single-element transducer in conjunction with Definity Microbubbles (10 μl/kg).
  Interventions: Device: Neuronavigation-guided single-element focused ultrasound transducer; Drug: Definity; Other: Magnetic Resonance Imaging (MRI) with or without gadolinium contrast agents; Other: Positron Emission Tomography (PET); Other: Amyvid

INTERVENTIONS:
Device: Neuronavigation-guided single-element focused ultrasound transducer — Non-invasive focused ultrasound-induced blood-brain barrier opening will be attempted using a single-element transducer, guided with a neuronavigation system.
Drug: Definity — Definity microbubbles (10 μl/kg) will be used in conjunction with the ultrasound transducer to temporarily open the blood brain barrier.
  Other Names: Perflutren Lipid Microsphere
Other: Magnetic Resonance Imaging (MRI) with or without gadolinium contrast agents — MRI scans will be completed at baseline and immediately after the focused ultrasound treatment to confirm BBB opening and safety. A follow-up MRI will be performed three days after treatment to confirm BBB closure, only in the case of successful BBB opening.
Other: Positron Emission Tomography (PET) — A follow-up PET scan will be performed three days after treatment to determine amyloid plaque load.
Other: Amyvid — To be used during the PET scan to determine uptake of Amyvid within the treated area.
  Other Names: 18F-Florbetapir

SUMMARY:
The purpose of this study is to test a new technique that may, in the future, help deliver medications to the brain of people with Alzheimer's disease. Participants in this study will undergo a focused ultrasound treatment to the brain, along with Magnetic Resonance Imagine (MRI) and Positron Emission Tomography (PET) scans.

DETAILED DESCRIPTION:
Central nervous system disorders are currently being symptomatically treated since the molecular events provoking their onset have not been yet identified. Drug delivery techniques have to overcome the almost impermeable blood-brain barrier (BBB) and can be grouped into two main categories: (i) invasive and targeted, and (ii) non-invasive and non-targeted methods. However, the technological advances of the past decades revealed the immense potential of focused ultrasound (FUS) in transcranial applications. In contrast to other techniques, FUS-mediated BBB opening is both non-invasive and targeted. The localized energy delivery coupled with the circulation of intravenously administered microbubbles initiates biological effects confined only to the vessel walls and contained only in the targeted region within the brain.

The purpose of the study is to assess the safety and feasibility of focused ultrasound-induced blood-brain barrier opening in Alzheimer's disease patients, using a single-element transducer with neuronavigation guidance. The investigators will also test whether treatment with focused ultrasound alone alters the amyloid protein levels in the treated brain areas and its potential effects on the cognitive function of Alzheimer's patients.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older.
* Diagnosis of early Alzheimer's disease (AD) or mild cognitive impairment (MCI) at minimum. All following criteria must be met:

  * Probable MCI or AD consistent with criteria outlined in (McKhann et al 2011, Petersen et al 2018).
  * Mini Mental State Examination (MMSE) score between 12 and 26.
  * Modified Hachinski Ischemia Scale (MHIS) score of <= 4
  * Short form Geriatric Depression Scale (GDS) score of <= 6.
  * PET scan confirming amyloid plaque load using Amyvid (18F-Florbetapir).
* Ability to provide informed consent.

Exclusion Criteria:

* Contraindication for Magnetic Resonance Imaging (MRI).
* Contra-indication history or hypersensitivity to MRI contrast agents (e.g., Dotarem) or microbubbles (e.g., Definity).
* Prior brain surgery, including deep brain stimulation.
* Metallic implants.
* Moderate or severe uncontrolled hypertension (systolic blood pressure > 140 mmHg).
* Abnormal coagulation profile, e.g. hemophilia A or B.
* Coagulopathy or under anticoagulant therapy.
* History of stroke or cardiovascular disease.
* Active/detectable gingivitis, herpes simplex, hepatitis, tuberculosis, and minor skin or respiratory infections.
* History of seizure disorder.
* History of asthma or allergies to food or medication with significant symptoms in past 3 years.
* Severe brain atrophy.
* Inability to comply with the procedures of the protocol, including follow-up MRI scans.
* Pregnancy or lactation.
* Impaired renal function with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 provided by a standard blood test at maximum 2 weeks prior to the ultrasound treatment.
* Active infection/inflammation.
* Acute or chronic hemorrhages, i.e. > 4 lobar microbleeds, and no siderosis or macrohemorrhages.
* Tumors or space occupying lesions.
* Meningeal enhancements.
* Intracranial hypotension.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Konofagou, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers.

REFERENCES:
- [Background] Wu SY, Aurup C, Sanchez CS, Grondin J, Zheng W, Kamimura H, Ferrera VP, Konofagou EE. Efficient Blood-Brain Barrier Opening in Primates with Neuronavigation-Guided Ultrasound and Real-Time Acoustic Mapping. Sci Rep. 2018 May 22;8(1):7978. doi: 10.1038/s41598-018-25904-9. PMID 29789530
- [Background] Pouliopoulos AN, Wu SY, Burgess MT, Karakatsani ME, Kamimura HAS, Konofagou EE. A Clinical System for Non-invasive Blood-Brain Barrier Opening Using a Neuronavigation-Guided Single-Element Focused Ultrasound Transducer. Ultrasound Med Biol. 2020 Jan;46(1):73-89. doi: 10.1016/j.ultrasmedbio.2019.09.010. Epub 2019 Oct 25. PMID 31668690
- [Derived] Karakatsani ME, Ji R, Murillo MF, Kugelman T, Kwon N, Lao YH, Liu K, Pouliopoulos AN, Honig LS, Duff KE, Konofagou EE. Focused ultrasound mitigates pathology and improves spatial memory in Alzheimer's mice and patients. Theranostics. 2023 Jul 14;13(12):4102-4120. doi: 10.7150/thno.79898. eCollection 2023. PMID 37554284
- [Derived] Mathew AS, Gorick CM, Price RJ. Multiple regression analysis of a comprehensive transcriptomic data assembly elucidates mechanically- and biochemically-driven responses to focused ultrasound blood-brain barrier disruption. Theranostics. 2021 Oct 11;11(20):9847-9858. doi: 10.7150/thno.65064. eCollection 2021. PMID 34815790
- See also: Ultrasound Elasticity Imaging Laboratory - Columbia University — https://ueil.bme.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Focused Ultrasound Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Focused Ultrasound Treatment
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
MMSE [Mean (Standard Deviation); unit: score on a scale] — The MMSE is a questionnaire that is used to measure cognitive impairment. The total score range is 0 to 30, with a higher score indicating a better outcome.
  score on a scale | 18.8 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Individuals With Successful Opening of the BBB
Description: The total number of individuals with successful opening of the BBB will be assessed. Blood-brain barrier opening volume will be measured in mm^3 through contrast-enhanced T1-weighted MRI on the day of the focused ultrasound treatment and 3 days after treatment, to confirm blood-brain barrier restoration.
Time Frame: Baseline through 3 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Focused Ultrasound Treatment
Number analyzed (Participants) | 6
Participants | 5

2. Primary Outcome: Total Number of Safety Events Related to Opening of BBB
Description: The total number of safety events related to opening of the BBB as assessed by T2 and susceptibility-weighted (SWI) MRI. Safety will be established by the presence and the total area of hyper-intense or hypo-intense areas in the T2 and SWI scans.
Time Frame: Baseline through 3 days post-treatment
Measure: Number; unit: adverse events
Arm/Group | Focused Ultrasound Treatment
Number analyzed (Participants) | 6
adverse events | 1

3. Secondary Outcome: Percent Change in Amyloid PET Signal Intensity
Description: Amyloid plaques will be assessed through PET imaging before and after the focused ultrasound treatment. The standardized uptake value ratio images (SUVr) will be compared before and after the FUS treatment, to investigate if there is a change in the uptake of 18F-Florbetapir within the treated area.
Time Frame: Screening through 3 weeks post-treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Focused Ultrasound Treatment
Number analyzed (Participants) | 6
percent change | -1.47 (0.77)

4. Secondary Outcome: Change in Mini-Mental State Examination (MMSE) Score
Description: The MMSE is a questionnaire that is used to measure cognitive impairment. The total score range is 0 to 30, with a higher score indicating a better outcome. Cognitive function will be assessed before and after the focused ultrasound treatment to determine the change in MMSE.
Time Frame: Screening through 3 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Focused Ultrasound Treatment
Number analyzed (Participants) | 6
score on a scale | -2.5 (2.93)

ADVERSE EVENTS:
Time Frame: Up to 5 months
Arm/Group | Focused Ultrasound Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Focused Ultrasound Treatment (N=6)
Mild focal edema (Injury, poisoning and procedural complications) | 1 (1) — Magnetic resonance imaging of one subject displayed a mild focal cortical and subcortical edema and superficial hemorrhage, likely meningeal. The subject was asymptomatic and the abnormalities resolved in the follow-up scans on day 15.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT04118764/Prot_SAP_000.pdf